CLINICAL TRIAL: NCT06285812
Title: OTO-MATIC: Otitis Treatment With OtoSight™ - Modification of Antibiotic Treatment Intervention in Children
Brief Title: Otitis Treatment With OtoSight™ - Modification of Antibiotic Treatment Intervention in Children
Acronym: OTO-MATIC
Status: Active, not recruiting | Type: Observational
Sponsor: PhotoniCare, Inc. (Industry)
Collaborators: TTi Health Research & Economics (Unknown)
Responsible Party: Sponsor
Other Study IDs: 000003
Record Dates: First submitted 2024-02-01; First posted 2024-02-29 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Otitis Media Acute
Keywords: Otitis Media with Effusion; Ear Infection; Optical Coherence Tomography; Otitis Media; Machine Learning
MeSH Terms: conditions — Otitis Media; Otitis Media with Effusion; Otitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Standard of Care #1: Prospective Randomized Control Trial (RCT)
- OtoSight #1: Prospective Randomized Control Trial (RCT)
  Interventions: Device: OtoSight Middle Ear Scope
- OtoSight #2: Case and provider match
  Interventions: Device: OtoSight Middle Ear Scope
- Standard of Care #2: Retrospective case and provider matched controls

INTERVENTIONS:
Device: OtoSight Middle Ear Scope — Subjects will be evaluated with the OtoSight Middle Ear Scope
  Groups: OtoSight #1; OtoSight #2

SUMMARY:
A pragmatic, mixed-method trial is to show the ability of OtoSight to change management of the pediatric patient presenting with ear pain in a way that improves patient outcomes and reduces costs.

DETAILED DESCRIPTION:
Mixed method, multi-center, pragmatic, cluster-randomized effectiveness-implementation investigation focused on pediatric subjects presenting with ear complaints at the office setting.

For the prospective randomized component, eligible clinicians at a given site will be randomized to one of two groups: the OtoSight intervention group or the usual care control group. There will be three (3) periods of post-intervention assessment: 10 days (optional), 6 months, and 12 months.

Eligible subjects will be automatically enrolled (or invited to enroll) in the clinical trial and will receive information. Because this is a non-interference design, frontline care clinicians randomized to either arm will be asked to: (1) assess the presence or absence of fluid in the middle ear; (2) record a diagnosis; and (3) treat the patient as they would according to the information available to them.

A separate retrospective historical matched control arm will also be conducted to analyze potential Hawthorne effect at a subset of collaborating practices or healthcare systems. Randomization of clinicians (and not children) will decrease contamination in the usual practice group (i.e., so clinicians are not asked to flip between intervention and usual care practices).

ELIGIBILITY:
For the Prospective Subjects

Inclusion Criteria:

* Pediatric subjects between 6 months and 17 years of age
* Pediatric subjects presenting for an office visit with ear-related pain (otalgia)/otic complaints/earache indicative of potential Otitis Media with Effusion (OME) or Acute Otitis Media (AOM)
* Pediatric subjects where otoscopy would traditionally be indicated
* Pediatric subjects whose parents or legally authorized representative (LAR) have signed an informed consent

Exclusion Criteria:

* The parent or guardian who attends visits does not speak the same language as their physician
* Pediatric subjects enrolled in another clinical trial
* Pediatric subjects with:
* Signs of severe chronic illness (e.g., immunodeficiency, congenital heart disease, encephalopathy, pulmonary disease other than asthma, and disorder of the ear, nose and throat) or any clinically significant illness or condition that, in the opinion of the investigator, would prohibit the subject from participating in the trial
* Anatomical conditions that would affect their ability to undergo an otoscopy.

For the Retrospective Case Match Controls

Inclusion Criteria:

* Pediatric subjects between 6 months and 17 years of age (< 18 years old).
* Index visit took place 11 - 25 months prior to the Treatment match's Baseline Visit.
* Index visit was for an ear-related chief complaint.
* An otoscopic exam was completed at index visit.
* Subjects have a follow up visits (telehealth included) in the time period between the index visit and firstTreatment subject's enrollment date.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Any pediatric patient between 6 months and 17 years of age scheduled for an office visit with ear-related complaints, deemed suitable for otoscopy assessment.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change the clinician rate of antibiotic prescriptions | Baseline to 12 month Follow Up
  Antibiotic stewardship
Change the number of antibiotic rounds per patient | Baseline to 12 month Follow Up
  Antibiotic stewardship
Change costs associated with management of pediatric patients presenting with ear-related pain | Baseline to 21 month Follow Up
  Change in overall costs

SECONDARY OUTCOMES:
Change in unnecessary antibiotic prescriptions | Baseline to 12 month Follow Up
  Change in unnecessary antibiotic prescriptions based on reported diagnosis and treatment recommendations of providers
Change in prescription adherence | Baseline to 12 month Follow Up
  Change in prescription adherence
Change in antibiotic prescription rate when fluid not present | Baseline to 12 month Follow Up
  Change in antibiotic prescriptions rate when fluid is not present based on reported treatment recommendations of providers
Improve patient outcomes | Baseline to 12 month Follow Up
  Change in progression to recurrent AOM (rAOM) based on tracking provider diagnoses
Change medical resource utilization | Baseline to 30 days Follow Up
  Change in follow-up visit frequency, ENT (Ear, Nose, and Throat) referral frequency
Change unnecessary medical intervention | Baseline to 12 month Follow Up
  Change in amount of unnecessary medical intervention (e.g., tympanostomy tube surgeries) based on tracking provider treatment recommendations and diagnoses
Impact clinician confidence | Baseline to 12 month Follow Up
  Change in clinician confidence scores reported on Provider CRF
Impact caregiver satisfaction | Baseline to 12 month Follow Up
  Change in clinician satisfaction scores reported on Provider CRF
Change in Health-related Quality of Life (HQoL) | Baseline to 12 month Follow Up
  Change in HQoL scores reported on the OMO-22 and OM-6

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Children's National Hospital, Washington D.C., District of Columbia
  - Abba Medical Group LLC, Miami, Florida
  - AdventHealth Children's Research, Orlando, Florida
  - Trillim Health, Rochester, New York
  - Cyn3rgy Research, Gresham, Oregon
  - Carolina ENT, Orangeburg, South Carolina
  - HealthStar Physicians, Morristown, Tennessee

IPD SHARING:
Plan to Share IPD: No